CLINICAL TRIAL: NCT01978561
Title: Pregnancy, Delivery, And Neonatal Outcomes In Subjects With Ongoing Pregnancies Established During Study NT-03 (Thrive-IVF Follow-Up)
Brief Title: Follow-Up Of Pregnancies Established During Study NT-03 (Thrive-IVF Follow-Up)
Acronym: Thrive-IVF F/U
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NT-04
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Repeated IVF Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Follow-Up after dosing with NT100 Dose 1 (Experimental): Follow-Up after dosing with NT100 Dose 1
  Interventions: Biological: Post dosing with NT100
- Follow-Up after dosing with NT100 Dose 2 (Experimental): Follow-Up after dosing with NT100 Dose 2
  Interventions: Biological: Post dosing with NT100
- Follow-Up after dosing with Placebo (Placebo Comparator): Follow-Up after dosing with Placebo
  Interventions: Other: Post dosing with Placebo

INTERVENTIONS:
Biological: Post dosing with NT100
  Arms: Follow-Up after dosing with NT100 Dose 1; Follow-Up after dosing with NT100 Dose 2
Other: Post dosing with Placebo
  Arms: Follow-Up after dosing with Placebo

SUMMARY:
The purpose of this study is to evaluate pregnancy, delivery, and neonatal outcomes in subjects who maintain ongoing clinical pregnancies through Week 10 of gestation in NT-03.

DETAILED DESCRIPTION:
NT-04 is a follow-up study that will include subjects who received at least one dose of study drug and maintain ongoing clinical pregnancies through Week 10 of gestation during NT-03. NT-04 does not involve the administration of study drug treatment.

In NT-03, subjects who achieve an ongoing clinical pregnancy at Week 8 of gestation will undergo a repeat transvaginal ultrasound (TVU) at Week 10 of gestation (4 weeks after last dose of study drug). Subjects who are pregnant at Week 10 of gestation will be enrolled in NT-04.

Subjects in NT-04 will be contacted by telephone every 6 to 8 weeks until Week 38 of gestation, at which time subjects will be contacted every two weeks until confirmation of delivery. Information about pregnancy status and use of prescription medications will be collected at these telephone interviews.

Between Weeks 18 and 22 of gestation, an obstetrical ultrasound will be performed.

Following delivery, additional information will be obtained, including pregnancy outcome, gestational age at delivery, etc. Standardized photographs will be taken as part of a newborn assessment.

ELIGIBILITY:
Inclusion Criteria:

* At least one dose of study drug administered in NT-03
* Ongoing clinical pregnancy at Week 10 of gestation
* Able and willing to enroll in NT-04

Exclusion Criteria:

• None

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of live births | Within approximately 7 months after NT-03

SECONDARY OUTCOMES:
Number of stillbirths | Within approximately 7 months after study NT-03
Number of spontaneous abortions (miscarriages) | Within approximately 7 months after study NT-03
Number of congenital anomalies | Up to 4 weeks after birth
Number of severe neonatal adverse events | Up to 4 weeks after birth

REFERENCES:
- See also: Study NT-03, Thrive-IVF Research Study — http://www.thriveivf.com